CLINICAL TRIAL: NCT06101966
Title: A Novel Predictive Model and Risk Stratification for Early Metastasis in Cervical Cancer Patients After Radiotherapy
Brief Title: A Predictive Model for Early Metastasis in Cervical Cancer Patients After Radiotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: prof.Sun
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cervical Cancer; Radiotherapy; Distant Metastasis; Prognostic Model; Risk Factor
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cervical cancer patients with radiotherapy: The overall dose should be more than 75 Gy. patients received surgery should be excluded.
  Interventions: Radiation: external pelvic beam radiotherapy (EBRT) followed by individualized high-dose-rate intracavitary brachytherapy (HDR-ICBT)

INTERVENTIONS:
Radiation: external pelvic beam radiotherapy (EBRT) followed by individualized high-dose-rate intracavitary brachytherapy (HDR-ICBT) — Radical RT consisted of external pelvic beam radiotherapy (EBRT) and individualized high-dose-rate intracavitary brachytherapy (HDR-ICBT).Cisplatin-based concurrent chemoradiotherapy (CCRT) was recommended for CC patients unless for economic status, age consideration and patients' desires.

SUMMARY:
This study aims to help to screen out appropriate cases for consolidation therapy and more intensive follow up.

DETAILED DESCRIPTION:
Some cervical cancer patients experienced distant metastasis quickly after receiving complete radiotherapy and have a worse prognosis. However, there were few studies focused on these patients and with early distant metastasis. It is significant to predictive and screen out cervial cancer patients with a high risk of early metastasis for more comprehensive treatments and follow-up plans

ELIGIBILITY:
Inclusion Criteria:

* patients confirmed as cervical cancer by biopsies and treated with radiotherapy were initially enrolled

Exclusion Criteria:

* (1) patients treated with surgery. (2) patient received incomplete treatment somewhere else. (3) patients with cancer history. (4) patients with pelvic surgery history. (5) patients without complete pre-treatment medical information. (6) patients with unfinished radical radiotherapy. (7) patients suffered from metastasis within 3 months after radiotherapy. (8) patients without complete 1-year follow-up materials

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cervical cancer patients recevied definitive radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Early distant metastases | 3-12months
  Early distant metastasis defines as metastasis occurrence between 3 -12 months after radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okazawa-Sakai M, Mabuchi S, Isohashi F, Kawashima A, Yokoi E, Ogawa K, Kimura T. Predictors of distant relapse in patients with FIGO stage IIB-IVA cervical cancer treated with definitive radiotherapy. J Obstet Gynaecol Res. 2017 Nov;43(11):1743-1750. doi: 10.1111/jog.13446. Epub 2017 Aug 17. PMID 28816403
- [Result] Liu X, Meng Q, Wang W, Zhou Z, Zhang F, Hu K. Predictors of Distant Metastasis in Patients with Cervical Cancer Treated with Definitive Radiotherapy. J Cancer. 2019 Jul 5;10(17):3967-3974. doi: 10.7150/jca.31538. eCollection 2019. PMID 31417641
- [Result] Li H, Wu X, Cheng X. Advances in diagnosis and treatment of metastatic cervical cancer. J Gynecol Oncol. 2016 Jul;27(4):e43. doi: 10.3802/jgo.2016.27.e43. PMID 27171673
- [Result] Zeng W, Huang L, Lin H, Pan R, Liu H, Wen J, Liang Y, Yang H. Development and Validation of a Nomogram for Predicting Postoperative Distant Metastasis in Patients with Cervical Cancer. Med Sci Monit. 2022 Apr 12;28:e933379. doi: 10.12659/MSM.933379. PMID 35410987